CLINICAL TRIAL: NCT05257577
Title: Factors Influencing Breast Cancer Resection Volumes And Their Impact on Treatment Outcome: a Prospective Multicenter Study (FIBRATIO)
Brief Title: Factors Influencing Breast Cancer Resection Volumes And Their Impact on Treatment Outcome (FIBRATIO)
Acronym: FIBRATIO
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Jyväskylä Central Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R21052
Record Dates: First submitted 2022-01-31; First posted 2022-02-25 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Quality of Life; Patient Satisfaction; Resection Margin; Surgical Margin; Multidisciplinary Communication
Keywords: breast conserving surgery; quality of life; resection margin; resection volume; reoperation rate
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction; Margins of Excision | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Breast conserving surgery
  Interventions: Procedure: Breast conserving surgery

INTERVENTIONS:
Procedure: Breast conserving surgery — Patients receive standard of care breast surgery and subsequent whole breast irradiation

SUMMARY:
The number of breast cancer survivors is constantly growing. Breast conserving surgery (BCS) is equal or superior to mastectomy both regarding survival and quality of life (QoL). Hence, as many patients as possible should be treated using BCS. The results indicate that the rate of mastectomies in Finland is higher than in Europe, while the rate of reoperations due to insufficient margins after BCS is lower in Finland than globally. With this study we aim to identify the optimal balance of radicality and tissue-conservation in BCS.

The aim of this study is to measure the volume of the resected breast tissue and the width of the healthy tissue margins and to compare these with the radiological and histological tumor size and with the size of the breast and their correlation with theoretically optimal and excised volumes.

This is a national prospective multicenter study conducted in five breast units. 250 women with primary, unilateral, cTis-T2 breast cancer eligible for BCS will be recruited. The diagnostics and treatment of the patients will be carried out following the Finnish national guideline. The size of the breast and the radiological size of the tumor will be measured preoperatively using mammograms and MRI. The histological tumor volume and the resection volume will be measured postoperatively. The optimal resection volume is calculated as the difference of the total resection volume and the volume of the tumor with an added 1 cm margin.

To map the impact of the treatment on QoL and body image, the patients are surveyed using EORTC-QLQ-C30 and BREAST-Q Breast Conserving Therapy Module QoL questionnaires preoperatively, 3-8 weeks postoperatively, and two years after the radiotherapy. Objective evaluation of the aesthetic outcome is assessed by the BCCT.core software that uses medical photographs taken at the same time points as the questionnaires are filled.

DETAILED DESCRIPTION:
1. Background

   Breast cancer is the most common cancer worldwide. The prognosis of early-stage breast cancer is good - more than 90 % of the patients are alive five years after diagnosis. Since many patients live decades after the diagnosis, besides oncological outcome, aesthetic, and functional outcomes are important for patients as a factor of quality of life (QoL) and global health. Breast conserving surgery (BCS) is equal or superior to mastectomy (Mx) both regarding survival and quality of life (QoL). Even if a patient has had immediate breast reconstruction their body image is inferior after mastectomy compared to those undergoing BCS.

   The aim of BCS is to remove the tumor with histologically negative margins defined as no ink on tumor for invasive carcinoma and 2 mm histological margin for ductal carcinoma in situ (DCIS). Wider negative margins do not improve local control when BCS is combined with radiotherapy (RT) but predispose patients to larger excision volumes and inferior cosmetic outcomes. Contrastingly, more conservative resections are associated with positive histological margins, which double the risk of tumor recurrence. Therefore, re-operation is performed for positive histological margins. Rates of re-excision vary widely between surgeons and facilities and according to recent international studies are up to 30 %. Re-operation is associated with several adverse outcomes such as delayed adjuvant treatment and impaired cosmetic outcomes and QoL.

   Finding the right balance between BCS and mastectomies, and the optimization of resection volumes are important considerations for surgical care of breast cancer. BCS rate and reoperation rate are both quality indicators of the European Society of Breast Cancer Specialists. The rate of mastectomies for early breast cancer in certified European breast units is approximately 25 %. There is no exact data on the rate of Mxs according to progression for Finland, however, it appears to be higher than in European units. Contrastingly, 8-13 % of the patients having BCS require a reoperation due to positive histological margins in Finland. These findings raise the question whether more BCS could be performed and with smaller macroscopic margins.

   Since the variation in reoperation rates, rates of mastectomies and resection volumes is largely unexplained, more research is needed to identify the root causes to enable effective interventions and raise the standards of care. Tumors and their anatomical location in the breast, breasts of the patients and surgical techniques vary and therefore measuring the BCS is challenging. Additionally, long-term cosmetic and functional outcomes are confounded by the effect of radiotherapy, and final outcome can be observed no earlier than two years after operation. In practice, measuring the ratio of the tumor volume to resection volume could provide comparable data and could even be a quality indicator of BCS. Our team has previously studied the technological innovations for intraoperative margin assessment and conducted retrospective analysis on the breast cancer margins in Finland. To effectively assess the factors affecting the resection volumes and obtained margins, a prospective approach is needed. A multicenter approach gives a comprehensive look on variation between institutions and surgeons. A study of this nature has not been conducted before.
2. Aim of the study

   The aim of this study is to measure the volume of the resected breast tissue and the width of the healthy tissue margins and to compare these with the radiological and histological tumor size and with the size of the breast and their correlation with theoretically optimal and excised volumes. These results help breast surgeons to find optimal balance of radicality and tissue-conservation.

   Primary endpoints
   * What is the effect of breast-related QoL and objective aesthetic outcome, as measured with BCCT.core, of the treatment on patient's overall QoL?
   * Are there differences in resection volumes and patient-related outcomes between surgeons or breast centers?
   * The ratio of theoretically optimal and excised resection volume for the tumor

   Secondary endpoints
   * What is the effect of radiotherapy on breast volume and shape?
   * What is the effect of the preoperative multidisciplinary team (MDT) treatment plan on the results?
   * What is the reoperation rate due to positive histological margins?
   * What is the effect of the tumor subtype, tumor size, DCIS component, tumor palpability or preoperative MRI imaging on the resection margins?
3. Research methods and execution

   3.1 Trial design and participants

   This is a national prospective multicenter study with a sample of 250 patients. The inclusion criterion is primary, unilateral cTis-T2 breast cancer eligible for BCS. Both conventional and volume-displacement oncoplastic techniques can be applied as long as the procedure is unilateral. The patients will be recruited from five Finnish breast units. For one surgeon at least 20 procedures are required. The sample size is powered to detect differences between centres and individual surgeons (alfa=0.05, beta=0.2, effect size 0.3) with the presumed loss of a maximum of 20% of patients at 2-year follow-up in terms of primary endpoints.

   Exclusion criteria for the study are metastatic, bilateral, and hereditary breast cancers or earlier breast cancer of the same or contralateral breast. Also, a symmetrisation procedure of the healthy breast simultaneously with the cancer operation or earlier breast procedures (excluding bilateral reduction mammoplasty/mastopexy) are contraindications. If the patient is not eligible for radiotherapy, has received neoadjuvant treatment, is pregnant or breastfeeding or is unable to provide an informed consent, she is not included in the study.

   For all patients the following data will be collected: age, BMI, comorbidity, smoking status, hormonal status, radiological data of the patient's breasts and the tumor, preoperative MDT data, histopathological data on the tumor and the margins, details of the operative treatment, postoperative complications, and details of the oncologic treatments.

   For all breast units the following characteristics will be collected: annual number of new primary breast cancers and primary breast cancer operations, Mx-rate, number of immediate and delayed breast reconstructions, number of surgeons, information about MDT principles For all breast surgeons the following characteristics will be collected: age, gender, specialty, years of work experience and workplace The diagnostics and treatment of the patients will be carried out following the Finnish national guideline, which is in line with international guidelines. The patients will not undergo any additional laboratory tests or imaging. The data will be collected from examinations done routinely during the diagnostic phase and follow-up phase.

   3.2 Volumetric measurements and the resection ratio

   The breast volume is calculated preoperatively and after radiotherapy by using mammography measurements (breast height, breast width and compression thickness) and the preoperative tumor volume by mammography and/or by the MRI. The effect of radiotherapy on breast size is calculated by comparing the preoperative and postoperative volume of the breast while considering the resection volume.

   The fresh surgical specimen is submerged in saline and its volume is measured using calculations based on Archimedes principle and Newton's third law. The radiological and histological tumor volume is calculated assuming the tumor to resemble an obloid spheroid.

   Optimal resection volume (ORV) is defined as the spherical volume of the tumor with an added 1.0 cm margin of healthy breast tissue. Total resection volume (TRV) is the measured volume of the fresh surgical specimen. TRV is compared to ORV to determine the excess of breast tissue resection (TRV/ORV=CRR) defined as calculated resection rate (CRR). Optimal CCR is 1.0.

   3.3 Quality of life and aesthetic results

   To map the impact of the treatment on QoL and body image, the patients are photographed and surveyed using QoL questionnaires (EORTC-QLQ-C30 version 3.0 and BREAST-Q Version 2.0 Breast Conserving Therapy Module) preoperatively, 3-8 weeks postoperatively and two years after the radiotherapy. Objective evaluation of the aesthetic outcome is assessed by the 'BCCT.core software' - INESC Porto Breast Research group based on medical photographs. The photographs are taken at same time points as QoL questionnaires are filled.

   The tumor-to-TRV ratios are analyzed between surgeons and centers while controlling for potential confounders at 3-8 weeks after surgery. Additionally, the correlation of the factors with aesthetic and QoL measures is analyzed at 3-8 weeks after surgery and 2 years after RT when the effect of radiation and adjuvant therapies is also fully included.
4. Schedule

The trial inclusion will begin in the spring 2022. Before the inclusion we will do a pilot study of five patients to validate the measuring techniques, the QoL questionnaires and the BCCT.core program.

The results will be analyzed at two time points:

1. 3-8 weeks after the operation
2. two years after the radiotherapy

The final results of the study should be available during 2025. The results will be published in peer-reviewed journals of surgical oncology.

ELIGIBILITY:
Inclusion Criteria:

* primary, solitary/multifocal, unilateral cTis-T2 breast cancer eligible for BCS
* DCIS, ductal, lobular and other subtypes of invasive breast cancer (excluding LCIS and ADH)
* ASA 1-2 and life expectancy more than 3 years
* mammogram done with a device showing compression thickness
* no previous breast surgery (bilateral reduction mammoplasty or mastopexy accepted)

Exclusion Criteria:

* metastatic breast cancer
* previous ipsi- or contralateral breast cancer
* bilateral breast cancer
* hereditary breast cancer
* contralateral symmetrization procedure in conjunction with the cancer surgery
* contraindication for radiotherapy
* neoadjuvant treatment
* pregnancy or breastfeeding
* inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological female
Study Population: Females ages 18 - 80 years of age scheduled to undergo breast conserving surgery and subsequent whole breast radiotherapy for unilateral DCIS or invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-05-28 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Breast-related quality of life assessed by EORTC QLQ-C30, BREAST-Q Version 2.0 Breast Conserving Therapy Module and BCCT.core | 2-3 years
  What is the effect of breast-related QoL and objective aesthetic outcome, as measured by two QoL questionnires and with BCCT.core, of the treatment on patient's overall QoL?
Differences in resection volumes (cm3) and patient reported outcomes between surgeons and breast units | 2 years
  Are there differences in resection volumes and patient-related outcomes between surgeons or breast centers?
Calculated resection rate | 2 months
  The ratio of theoretically optimal and excised resection volume for the tumor

SECONDARY OUTCOMES:
Radiotherapy effects on the breast assessed by bilateral breast volume measurement by mammogram, and by BCCT.core | 2-3 years
  What is the effect of radiotherapy on breast volume and shape? Breast volume is measured preoperatively and two years after the radiotherapy. Breast volume based on mammogram data calculated using the formula proposed by Kalbhen et al, Am JRoentgenol. 1999: Volume = (π/4) × Breast height × Breast width × Compression thickness in cranio-caudal mammogram. Breast shape is assessed by BCCT.core.
Significance of the multidisciplinary team treatment plan on treatment outcome | 2-3 years
  What is the effect of the preoperative multidisciplinary team (MDT) treatment plan on the results? MDT planning will be assessed as YES or NO scale.
Reoperation rate | 1-7 months
  What is the reoperation rate due to positive histological margins?
Effect of the tumor subtype, tumor size, DCIS component, tumor palpability or preoperative MRI imaging on the resection margins? | 2 months
  What is the effect of the tumor subtype, tumor size, DCIS component, tumor palpability or preoperative MRI imaging on the resection margins?

CONTACTS AND LOCATIONS:
Overall Officials: Niku KJ Oksala, Professor, Principal Investigator — Tampere University Hospital, Tampere University
Locations (4):
- Finland (4):
  - Hospital Nova of Central Finland, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Agarwal S, Pappas L, Neumayer L, Kokeny K, Agarwal J. Effect of breast conservation therapy vs mastectomy on disease-specific survival for early-stage breast cancer. JAMA Surg. 2014 Mar;149(3):267-74. doi: 10.1001/jamasurg.2013.3049. PMID 24429935
- [Background] Waljee JF, Hu ES, Ubel PA, Smith DM, Newman LA, Alderman AK. Effect of esthetic outcome after breast-conserving surgery on psychosocial functioning and quality of life. J Clin Oncol. 2008 Jul 10;26(20):3331-7. doi: 10.1200/JCO.2007.13.1375. PMID 18612149
- [Background] Kelsall JE, McCulley SJ, Brock L, Akerlund MTE, Macmillan RD. Comparing oncoplastic breast conserving surgery with mastectomy and immediate breast reconstruction: Case-matched patient reported outcomes. J Plast Reconstr Aesthet Surg. 2017 Oct;70(10):1377-1385. doi: 10.1016/j.bjps.2017.05.009. Epub 2017 May 18. PMID 28712883
- [Background] Cardoso F, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rubio IT, Zackrisson S, Senkus E; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Early breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-updagger. Ann Oncol. 2019 Aug 1;30(8):1194-1220. doi: 10.1093/annonc/mdz173. No abstract available. PMID 31161190
- [Background] Volders JH, Negenborn VL, Haloua MH, Krekel NMA, Jozwiak K, Meijer S, M van den Tol P. Cosmetic outcome and quality of life are inextricably linked in breast-conserving therapy. J Surg Oncol. 2017 Jun;115(8):941-948. doi: 10.1002/jso.24615. Epub 2017 Mar 23. PMID 28334419
- [Background] Valero MG, Mallory MA, Losk K, Tukenmez M, Hwang J, Camuso K, Bunnell C, King T, Golshan M. Surgeon Variability and Factors Predicting for Reoperation Following Breast-Conserving Surgery. Ann Surg Oncol. 2018 Sep;25(9):2573-2578. doi: 10.1245/s10434-018-6526-2. Epub 2018 May 21. PMID 29786129
- [Background] van Leeuwen MT, Falster MO, Vajdic CM, Crowe PJ, Lujic S, Klaes E, Jorm L, Sedrakyan A. Reoperation after breast-conserving surgery for cancer in Australia: statewide cohort study of linked hospital data. BMJ Open. 2018 Apr 10;8(4):e020858. doi: 10.1136/bmjopen-2017-020858. PMID 29643165
- [Background] Biganzoli L, Marotti L, Hart CD, Cataliotti L, Cutuli B, Kuhn T, Mansel RE, Ponti A, Poortmans P, Regitnig P, van der Hage JA, Wengstrom Y, Rosselli Del Turco M. Quality indicators in breast cancer care: An update from the EUSOMA working group. Eur J Cancer. 2017 Nov;86:59-81. doi: 10.1016/j.ejca.2017.08.017. Epub 2017 Sep 28. PMID 28963914
- [Background] Garcia-Etienne CA, Tomatis M, Heil J, Friedrichs K, Kreienberg R, Denk A, Kiechle M, Lorenz-Salehi F, Kimmig R, Emons G, Danaei M, Heyl V, Heindrichs U, Rageth CJ, Janni W, Marotti L, del Turco MR, Ponti A; eusomaDB Working Group. Mastectomy trends for early-stage breast cancer: a report from the EUSOMA multi-institutional European database. Eur J Cancer. 2012 Sep;48(13):1947-56. doi: 10.1016/j.ejca.2012.03.008. Epub 2012 Apr 4. PMID 22483323
- [Background] Ojala K, Meretoja TJ, Mattson J, Salminen-Peltola P, Leutola S, Berggren M, Leidenius MH. The quality of preoperative diagnostics and surgery and their impact on delays in breast cancer treatment - A population based study. Breast. 2016 Apr;26:80-6. doi: 10.1016/j.breast.2015.12.009. Epub 2016 Feb 1. PMID 27017246
- [Background] Niinikoski L, Leidenius MHK, Vaara P, Voynov A, Heikkila P, Mattson J, Meretoja TJ. Resection margins and local recurrences in breast cancer: Comparison between conventional and oncoplastic breast conserving surgery. Eur J Surg Oncol. 2019 Jun;45(6):976-982. doi: 10.1016/j.ejso.2019.02.010. Epub 2019 Feb 11. PMID 30795953
- [Background] Lepomaki M, Karhunen-Enckell U, Tuominen J, Kronqvist P, Oksala N, Murtola T, Roine A. Tumor margins that lead to reoperation in breast cancer: A retrospective register study of 4,489 patients. J Surg Oncol. 2022 Mar;125(4):577-588. doi: 10.1002/jso.26749. Epub 2021 Nov 15. PMID 34779520
- [Background] Sutinen M, Kontunen A, Karjalainen M, Kiiski J, Hannus J, Tolonen T, Roine A, Oksala N. Identification of breast tumors from diathermy smoke by differential ion mobility spectrometry. Eur J Surg Oncol. 2019 Feb;45(2):141-146. doi: 10.1016/j.ejso.2018.09.005. Epub 2018 Oct 15. PMID 30366874
- [Background] Kontunen A, Karhunen-Enckell et al. Tissue Identification From Surgical Smoke by Differential Mobility Spectrometry: An in Vivo Study. IEEE Access 2021; 9:168355-168367. DOI 10.1109/ACCESS.2021.3136719
- [Background] Lagendijk M, Vos EL, Ramlakhan KP, Verhoef C, Koning AHJ, van Lankeren W, Koppert LB. Breast and Tumour Volume Measurements in Breast Cancer Patients Using 3-D Automated Breast Volume Scanner Images. World J Surg. 2018 Jul;42(7):2087-2093. doi: 10.1007/s00268-017-4432-6. PMID 29299647
- [Background] Fujiwara T, Yano K, Tanji Y, Hosokawa K. Simple and accurate volume measurement of mastectomy specimens. Eur J Plast Surg. 36:275-276, 2013
- [Background] Krekel N, Zonderhuis B, Muller S, Bril H, van Slooten HJ, de Lange de Klerk E, van den Tol P, Meijer S. Excessive resections in breast-conserving surgery: a retrospective multicentre study. Breast J. 2011 Nov-Dec;17(6):602-9. doi: 10.1111/j.1524-4741.2011.01198.x. PMID 22050281
- [Background] Cardoso MJ, Cardoso JS, Vrieling C, Macmillan D, Rainsbury D, Heil J, Hau E, Keshtgar M. Recommendations for the aesthetic evaluation of breast cancer conservative treatment. Breast Cancer Res Treat. 2012 Oct;135(3):629-37. doi: 10.1007/s10549-012-1978-8. Epub 2012 Feb 4. PMID 22307267
- [Background] Kalbhen CL, McGill JJ, Fendley PM, Corrigan KW, Angelats J. Mammographic determination of breast volume: comparing different methods. AJR Am J Roentgenol. 1999 Dec;173(6):1643-9. doi: 10.2214/ajr.173.6.10584814.